

\*\*FOR CCI USE ONLY\*\*

Approved by the Beth Israel Deaconess Medical Center Committee on Clinical Investigations:

Consent Approval Date: 04/23/2019

Protocol Number: 2018P000040



# INFORMED CONSENT FORM TO TAKE PART IN A RESEARCH STUDY

SUBJECT'S NAME:

TITLE OF RESEARCH PROTOCOL: EEG changes with meditation: A proposal to analyze EEG

changes with a simple, online, guided meditative tool

PRINCIPAL INVESTIGATOR: Balachundhar Subramaniam, MD, MPH

**PROTOCOL NUMBER:** 

## **INTRODUCTION:**

- This is a research study;
- Your participation is voluntary;
- A research study includes only people who choose to take part;
- You may or may not benefit from participating in the study. However, your participation may help others in the future as a result of knowledge gained from the research;
- You may leave the study at any time;
- ➤ If you choose not to take part, or if you leave the study, your decision will in no way harm your relationship with any member of the research team or any other individuals at Beth Israel Deaconess Medical Center.

Please read this consent form carefully and ask the investigators or study staff to explain any words or information that you do not clearly understand. Once you read this consent form and understand what your participation in this study will involve, you will be asked to sign this form if you wish to take part. You will be given a signed copy of the form to keep for your records.

## DISCLOSURE OF SPECIAL INTERESTS OF BIDMC AND INVESTIGATORS

This study is being conducted by Balachundhar Subramaniam MD, MPH. There is no funding agency in this study. Neither BIDMC nor Dr. Subramaniam has/have any additional interests in this research project. The PI is an unpaid consultant to the Isha foundation. Isha Foundation is a volunteer-based, non-profit organization that serves as a resource for yoga science and meditation.

## WHOM TO CONTACT IF YOU HAVE QUESTIONS OR PROBLEMS

If you have any questions, concerns or complaints about this research or experience any problems, you should contact Balachundhar Subramaniam MD, MPH at [617] 754-2675.



TITLE OF RESEARCH PROTOCOL: **EEG changes with meditation:** A proposal to analyze **EEG changes with a simple, online,** guided meditative tool

PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam,

MD, MPH

PROTOCOL #: 2018P000040



## **PURPOSE**

The purpose of this study is to understand how meditation may affect EEG patterns in the brain. An electroencephalogram (EEG) is a test that measures the brain's electrical activity. This involves placing a cap with small, flat metal discs (electrodes) on your head. Your brain cells communicate via electrical impulses and are active all the time, even when you're asleep. This activity shows up as wavy lines on an EEG recording.

# STUDY PARTICIPANTS

You have been asked to be in the study because you are a healthy volunteer. Approximately 15 people will take part in this study at Beth Israel Deaconess Medical Center.

## **DESCRIPTION OF STUDY DETAILS**

If you agree to be in this study, you will be asked to read and sign this consent form. After you sign the consent form and you qualify to take part in this research study, the following things will happen:

- 1. Based on your experience with meditation, you will be placed into one of two groups:
  - a) Novice meditator: No meditation practice in the previous year and < 20 entire lifetime hours
  - b) Expert meditator: Meditation ≥ 30 minutes per day for at least 5 days per week over the past 1 year

## 2. Research Procedures:

## Introduction to meditation

The research team will give you an introduction to Isha Kriya (IK) meditation, along with written instructions. It is a meditation using thought and mindful breathing that can be learned quickly. It does not incorporate a spiritual or religious focus.

# EEG monitored meditation sessions

While undergoing real time EEG monitoring, you will be asked to perform simple exercises and to meditate. We will ask you to undergo 2 EEGs: one at the beginning of the study and another approximately 6 weeks later. Each session should take approximately 1 hour.

## Daily meditation

During the 6 weeks between the EEGs, you will be asked to meditate two (2) times each day for approximately 12 minutes each time. You will also be given a Meditation Diary to track your meditation sessions. During this time, the research team may contact you via telephone



TITLE OF RESEARCH PROTOCOL: **EEG changes with meditation:** A proposal to analyze EEG changes with a simple, online, guided meditative tool

PRINCIPAL INVESTIGATOR'S NAME: **Balachundhar Subramaniam**, **MD**, **MPH** 

PROTOCOL #: 2018P000040

to answer any questions.



# **RISKS AND DISCOMFORTS**

As a result of your participation in this study, you are at risk for side effects listed in this section. You should discuss these with the investigator and with your regular doctor if you choose.

## EEG:

Noninvasive EEG monitoring is considered a safe procedure. It has no discomfort and produces no sensation. In addition, there is no risk of electric shock. EEG will be performed by trained study staff.

## Meditation:

The meditation intervention only involves thought and mindful breathing. We do not anticipate any physical risk.

## LOSS OF CONFIDENTIALITY

There is the potential for loss of confidentiality by participating in this study. Every effort will be made to protect the confidentiality of your identifiable information.

However, if your participation becomes known, it could create a problem or hardship for you depending upon the type of information disclosed. In some situations, it is possible that you would be placed at risk for damage to your health care, professional standing or ability to get access to health or other insurance. We take your privacy very seriously, and will be following a very careful plan to keep all your information confidential.

### CONFIDENTIALITY

Information learned from your participation in this study and from your medical record may be reviewed and photocopied by the Food and Drug Administration (FDA) and/or other federal and state regulatory agencies, and by accreditation agencies, the Committee on Clinical Investigations, the Human Subjects Protection Office and others involved in research administration of the Beth Israel Deaconess Medical Center with protection of confidentiality so far as permitted by applicable law. Information resulting from this study and from your medical record may be used for research purposes and may be published; however, you will not be identified by name in such publications.

# **POSSIBLE BENEFITS**

There is no direct benefit to you from being in this study. However, your participation may help others in the future as a result of knowledge gained from the research.

# OTHER AVAILABLE OPTIONS

Taking part in this study is voluntary. Instead of being in this study, you have the option of not enrolling in the study.



TITLE OF RESEARCH PROTOCOL: **EEG changes with meditation:** A proposal to analyze **EEG changes with a simple, online,** guided meditative tool

PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam,

MD, MPH

PROTOCOL #: 2018P000040



## IF YOU DECIDE NOT TO TAKE PART IN THE STUDY

Participation in this study is voluntary. You have the right to decide not to take part in this study. If you choose to participate, you have the right to leave the study at any time. Your decision to not participate will not result in any penalties or loss of benefits to you. The investigators will tell you about new information that may affect your willingness to stay in this study.

If you decide not to participate in the study or decide to leave the study early, your decision will not affect your relationship with the research team or any other individual at Beth Israel Deaconess Medical Center.

# INVESTIGATORS RIGHT TO STOP THE STUDY

The investigators have the right to end your participation in this study if they determine that you no longer qualify to take part, or if it would be dangerous for you to continue, or if you do not follow study procedures as directed by the investigators. Beth Israel Deaconess Medical Center or the funding source may stop the study at any time.

### COSTS AND/OR PAYMENTS TO YOU

# **COSTS COVERED BY STUDY**

You will not be charged for the EEG monitoring that is a part of this research study.

# PAYMENTS TO YOU:

You will not be paid for participating in the study. However, you will receive a voucher to cover parking costs at the BIDMC parking garage each time you come for an EEG.

# OTHER IMPORTANT INFORMATION

A description of this clinical trial will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a> as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# AUTHORIZATION FOR USE AND DISCLOSURE OF YOUR PROTECTED HEALTH INFORMATION

As part of this study, we will be collecting, using and sharing with others information about you. Please review this section carefully as it contains information about the federal privacy rules and the use and disclosure of your information.

# PROTECTED HEALTH INFORMATION [PHI]

By signing this informed consent document, you are allowing the investigators and other authorized



TITLE OF RESEARCH PROTOCOL: **EEG changes with meditation:** A proposal to analyze EEG changes with a simple, online, guided meditative tool

PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam,

MD, MPH

PROTOCOL#: 2018P000040



personnel to use [internally at BIDMC] and disclose [to people and organizations outside the BIDMC workforce identified in this consent] health information about you. This may include information about you that already exists (for example: your medical records and other sources of health information, demographic information, the results of any laboratory tests, and mental health records if applicable) as well as any new information generated as part of this study. This is your Protected Health Information.

People/Groups at BIDMC Who Will Share and Use Your Protected Health Information
Your Protected Health Information may be shared with and used by investigators working on this
study, including the supporting research team (such as research assistants and coordinators,
statisticians, data managers, laboratory personnel, pharmacy personnel, and administrative
assistants), and may also be shared and used by other health care providers at BIDMC who have
treated you in the past and have information relevant to the research, or who provide services to you
in connection with the research. Your Protected Health Information may also be shared with the
members and staff of the Committee on Clinical Investigations of Beth Israel Deaconess Medical
Center, which is responsible for reviewing studies for the protection of the research subjects.

# PEOPLE/GROUPS OUTSIDE OF BIDMC WITH WHOM YOUR PROTECTED HEALTH INFORMATION WILL BE SHARED

We will take care to maintain confidentiality and privacy about you and your Protected Health Information. We may share your Protected Health Information with the following groups so that they may carry out their duties related to this study:

- The Food and Drug Administration [FDA], the Department of Health and Human Services [DHHS], the National Institute of Health [NIH], the Office for Human Research Protections [OHRP], and other federal and state agencies that may have jurisdiction over the research
- Hospital and Clinical Research Accrediting Agencies
- Research groups not affiliated with BIDMC that are involved in analyzing data related to the research

Those who receive your Protected Health Information during the course of the research may not be required by the federal privacy regulations to protect it, and they may make further disclosures to others and use your information without being subject to penalties under those laws.

# WHY WE ARE USING AND SHARING YOUR PROTECTED HEALTH INFORMATION

The main reason for using and sharing your Protected Health Information is to conduct and oversee the research as described in this Informed Consent Document. There are many other reasons beyond the research for which BIDMC may use or disclose your Protected Health Information. Not all of these reasons require your express written authorization. For example, we will use and share



TITLE OF RESEARCH PROTOCOL: **EEG changes with meditation:** A proposal to analyze **EEG changes with a simple, online,** guided meditative tool

PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam,

MD, MPH

PROTOCOL#: 2018P000040



your Protected Health Information to ensure that the research meets legal, institutional and accreditation requirements and to conduct public health activities. The various ways in which BIDMC may use and disclose your protected health information without your authorization are explained in a document called the Notice of Privacy Practices. If you have not received a copy of BIDMC's Notice of Privacy Practices, please ask us for one and review it before signing this form. In addition to signing this document, you may also be asked to sign a BIDMC General Agreement form acknowledging that you have received the BIDMC Notice of Privacy Practices.

## No Expiration Date - Right to Withdraw Authorization

Your authorization for the use and disclosure of your Protected Health Information in this Study shall never expire. However, you may withdraw your authorization for the use and disclosure of your Protected Health Information at any time provided you notify the Principal Investigator in writing. If you would like to take back your authorization so that your Protected Health Information can no longer be used in this study, please send a letter notifying the Principal Investigator of your withdrawal of your authorization to Dr. Balachundhar Subramaniam at One Deaconess Road, CC 657, Beth Israel Deaconess Medical Center, Boston, MA 02215. Please be aware that the investigators in this study will not be required to destroy or retrieve any of your Protected Health Information that has already been used or disclosed before the Principal Investigator receives your letter, and they are permitted to continue to use and disclose your previously collected information as necessary to complete the research.

## **REFUSAL TO SIGN**

Your clinical treatment may not be conditioned upon whether you sign the Authorization for Research. However, if you choose not to sign this informed consent document and authorization for the use and disclosure of your Protected Health Information, you will not be allowed to take part in the research study.

#### RIGHT TO ACCESS AND COPY YOUR PHI

If you wish to review or copy your Protected Health Information as it is made part of your medical record, you may do so after the completion or termination of the study by sending a letter to the Principal Investigator requesting a copy of your Protected Health Information. You may not be allowed to inspect or copy your Protected Health Information until this study is completed or terminated.

## ADDITIONAL CONTACT FOR QUESTIONS OR CONCERNS

You may contact the Human Subjects Protection Office at [617] 975-8500 in the event that you would like to obtain information or to offer input about the research study. This office is independent of the investigator or investigator's research staff and can also assist with questions



TITLE OF RESEARCH PROTOCOL: **EEG changes with meditation:** A proposal to analyze **EEG changes with a simple, online,** guided meditative tool

PRINCIPAL INVESTIGATOR'S NAME: **Balachundhar Subramaniam**, **MD**, **MPH** 

PROTOCOL#: 2018P000040



relating to your rights as a participant in research, which may include questions, concerns or complaints about your participation in the study.



| Beth Israel Deaconess Medical Center | [CCI] Committee on Clinical Investigations<br>Page 8 of 9 |
|---|---|
| SUBJECT'S NAME: | SRAEL DEACON |
| TITLE OF RESEARCH PROTOCOL: <b>EEG changes with meditation:</b> | APPROVED BY THE |
| A proposal to analyze EEG changes with a simple, online, guided meditative tool | 04/22/2020 |
| PRINCIPAL INVESTIGATOR'S NAME: <b>Balachundhar Subramaniam</b> , <b>MD</b> , <b>MPH</b> | APPROVAL EXPIRATION DATE |
| PROTOCOL #: 2018P000040 | - CAL CE. |
| CONSENT FORM FOR CLINICAL RESEARCH I have read the previous page[s] of the consent form and the investigated study. I understand that I am free to ask additional questions. If I wish additional information regarding this research and my rights as | s a research subject, or if I believe I |
| have been harmed by this study, I may contact the Human Subjects Pr<br>I am aware that this is a research project and that unforeseen side effe | , |
| I understand that the Beth Israel Deaconess Medical Center has no for patients for medical injuries arising from this research. Medical treatm usual charge to me or to my insurer unless payment is otherwise provided in the control of the control | rmal program for compensating<br>ent will be provided for injuries at the |
| I understand that participation in this study is voluntary and I may refus<br>participation at any time without penalty, loss of benefits, or prejudice t<br>receive. | |
| I acknowledge that no guarantees have been made to me regarding the this study, and I consent to participate in the study and have been give | |
| Signature of Subject or Date Legally Authorized Representative | |

S (Parent if the subject is a minor) Relationship of Legally Authorized Representative to Subject The subject has been given the opportunity to read this consent form and to ask questions before signing, and has been given a copy. SIGNATURE OF INVESTIGATOR/Co-Investigator DATE PRINT INVESTIGATOR'S/Co-Investigator's NAME A signing co-investigator must be listed on the study's approved Research Staffing Form at the time of consent.



| * | Without Cities |
|---|---|
| | SUBJECT'S NAME: |
| | TITLE OF RESEARCH PROTOCOL: <b>EEG changes with meditation:</b> A proposal to analyze EEG changes with a simple, online, guided meditative tool |
| | PRINCIPAL INVESTIGATOR'S NAME: Balachundhar Subramaniam, MD, MPH |
| | PROTOCOL #: 2018P000040 |
| HE FOLLOWING SECTIONS ARE NOT NEEDED FOR ALL STU | |



#### UDIES AND SHOULD BE TH **UTILIZED AS INDICATED:**

If the subject is able to speak and understand English but is not able to read or write

| If the Subject is able to speak and understand English but is not able to read of write |
|---|
| I was present during the entire oral presentation of the informed consent and witnessed the subject's agreement to participate in the study. |
| Signature of Witness: |
| Printed Name of Witness: |
| Date: ——— |
| If the subject is able to understand English but is not physically able to read or write or see |
| I was present during the entire oral presentation of the informed consent and witnessed the subject's agreement to participate in the study. |
| Signature of Witness: |
| Printed Name of Witness: |
| Date: |
| If the subject is not English speaking and signed the translated Short Form in lieu of the English consent document. |
| As someone who understands both English and the language spoken by the subject, I interpreted, in the subject's language, the researcher's presentation of the English consent form. The subject was given the opportunity to ask questions. |
| Signature of Interpreter: |
| Printed name of Interpreter: |
| Date: |